CLINICAL TRIAL: NCT06134752
Title: Electroporation for Treatment of Persistent and Longstanding Persistent Atrial Fibrillation
Brief Title: Electroporation for Treatment of Atrial Fibrillation
Acronym: ELECTROAF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELECTROAF
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; pulse field ablation; radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation (Active Comparator): Pulmonary vein and left atrial posterior wall isolation with point by point radiofrequency ablation.
  Interventions: Other: Radiofrequency ablation
- Pulse field ablation (Experimental): Pulmonary vein and left atrial posterior wall isolation with point by point pulse field ablation.
  Interventions: Other: Pulse field ablation

INTERVENTIONS:
Other: Pulse field ablation — Point by point isolation of pulmonary veins and left atrial posterior wall
  Arms: Pulse field ablation
Other: Radiofrequency ablation — Point by point isolation of pulmonary veins and left atrial posterior wall
  Arms: Radiofrequency ablation

SUMMARY:
Comparison of pulmonary vein and left atrial posterior wall isolation durability and clinical outcome between radiofrequency and pulse field ablation in patients with persistent and longstanding persistent atrial fibrillation.

DETAILED DESCRIPTION:
Patients with persistent and longstanding persistent atrial fibrillation will be randomized to control and investigational group.

In control group they will receive pulmonary vein and posterior wall ("box lesion") isolation with point by point radiofrequency ablation utilizing the CLOSE protocol with predetermined interlesion distance of up to 6 mm and predetermined ablation index/lesion size index.

In investigational group they will receive pulmonary vein and posterior wall ("box lesion" and additional ablations inside the "box") isolation with point by point pulse field ablation with a predetermined interlesion distance of up to 6 mm and predetermined energy delivery settings.

30 minutes after the last ablation point a high-density mapping of the left atrium will be performed.

Preprocedurally all patients will undergo computer tomography angiography of the left atrium, which will be processed resulting in a three dimensional anatomy reconstruction that will be utilized during the procedures in conjunction with the three dimensional mapping system. Also, left atrial wall thickness will be determined and displayed on the three dimensional anatomy reconstruction.

Before and after radiofrequency and pulse field ablation a five minute bipolar and unipolar intracardiac electrogram recording will be performed at at least two predetermined locations according to wall thickness (at the thinest and at the thickest part of the wall) for later analysis of changes due to different modes of ablation with correlation to lesion durability at a three month re-mapping procedure.

Collection of full blood before and 24 and 48 hours after the procedure to analyse activation of inflammation, coagulation, and also nevral tissue injury and endotelial injury due to ablation. Deviation of markers from the baseline value before the procedure will serve as a measure of activation. Markers analysed: troponin (ng/ml), D dimer (mg/l fibrinogen equivalent units), protein S100 (ng/ml), protein NSE (ng/ml), NT proBNP (pg/ml), high sensitivity CRP (mg/l), interleukin (IL) 6 (pg/ml), procalcitonin (ng/ml), fibrinogen (g/l), P selectin /pg/ml).

Postprocedurally pateints will undergo a remapping procedure three months later to determine pulmonary vein and left atrial posterior wall isolation durability.

Pateints will be followed up with clinical checkup and 1-7 day ECG holters at 3, 6, 12 months.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation recorded with 12-lead ECG, holter ECG or implantable device on two occasions at least one week apart

Exclusion Criteria:

* history of previous catheter ablation, history of previous heart surgery, life expectancy less than one year, any lifethreatening severe acute condition, acute deep venous thrombosis, presence of intracardiac masses or thrombi.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Durability of isolation | 3 months
  Testing for durability of pulmonary vein and left atrial posterior wall isolation in both study arms with high density endocardial remapping.
  Absence of electrical activity or voltage inside ablation lines of less than 0.05 mV or presence of exit block upon pacing with local capture will be considered as proof of pulmonary vein and posterior left atrial wall isolation.

SECONDARY OUTCOMES:
Freedom from atrial arrhythmias | 12 months
  Freedom from atrial tachycardia, atrial flutter and atrial fibrillation during the follow up as assessed with 12-lead ECG and 1-7 day holter ECG recordings at 3, 6, 12 months. With holter recordings any arrhythmia lasting at least 30 seconds will be considered as a recurrence.
Intracardiac electrograms analysis | 1 day
  Five minute recording of bipolar and unipolar intracardiac electrograms with a high density mapping catheter at predetermined locations in pulmonary vein antra and left atrial posterior wall before and after radiofrequency and pulse field ablation at the index procedure. Offline analysis of recorded signals and correlation of immediate changes with persistence of durable lesions (isolation) or conduction gaps.
Recording of complications | 30 days
  Postprocedural endoscopy of the esophagus and endoscopic ultrasound of the esophagus up to 72 hours after the procedure for detection of esophageal injury. Recording of any intra and postprocedural complications up to a 30 day period.

CONTACTS AND LOCATIONS:
Overall Officials: Jernej Štublar, BSE, Study Chair — University Medical Centre Ljubljana
Locations (1):
- Cardiovascular Surgery Department, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No